CLINICAL TRIAL: NCT04298450
Title: ED to EPI: Using SMS (Text) Messaging to Improve the Transition from the Emergency Department to Early Psychosis Intervention for Young People with Psychosis
Brief Title: ED to EPI: Using SMS to Improve the Transition from the Emergency Department to Early Psychosis Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Institute for Clinical Evaluative Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 088/2019
Record Dates: First submitted 2020-03-03; First posted 2020-03-06 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-03

CONDITIONS: First Episode Psychosis; Psychosis; Psychotic Episode; Psychoses, Affective; Bipolar Disorder; Depressive Psychosis; Schizoaffective Disorder; Schizophreniform Disorders; Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Substance Induced Psychoses
Keywords: Early Psychosis Intervention; Mobile Health Intervention; Patient and Family Engagement; Pragmatic Clinical Trials; Transitions in Care
MeSH Terms: conditions — Psychotic Disorders; Affective Disorders, Psychotic; Bipolar Disorder; Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Psychoses, Substance-Induced

STUDY DESIGN:
Intervention Model Description: Immediately after study enrollment, participants will be randomized using an electronic data management system to the active or sham intervention. Randomization will be stratified by sex and referral source (main emergency department vs. Bridging Clinic vs. inpatient unit), using a computer algorithm to perform a blocked randomization assignment within strata.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will not be notified of treatment assignment, but based on the nature of the intervention, they cannot be fully masked. Their care provider may know treatment assignment if disclosed by the participant, or if they get notified that the participant is in distress. Treatment assignment will be known by the research personnel involved in managing the intervention and the database linking participant information to study identification numbers. Treatment assignment may be known by a co-principal investigator providing clinical supervision for adverse or serious events. Research personnel involved in qualitative interviews will also be aware of treatment assignment since only individuals receiving the active treatment participate. The lead principal investigator and research personnel involved in the chart review (where the primary outcome will be extracted) and other analyses will be masked to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active SMS Intervention (Experimental): Participants assigned to the experimental arm will receive the active SMS intervention. Participants in the active intervention group who consent to participate will be asked to complete a web-based survey. Based on survey findings, purposive sampling will be used to select a subsample of 12 to 20 participants for qualitative interviews.
  Interventions: Behavioral: Active SMS Intervention
- Sham SMS (Sham Comparator): Participants assigned to the sham comparator will receive the sham SMS intervention. They will not be re-contacted.
  Interventions: Behavioral: Sham SMS

INTERVENTIONS:
Behavioral: Active SMS Intervention — Welcome message letting participant know they will be contacted to book an appointment, followed by appointment reminders and other clinic information, psychoeducational materials, and a distress check-in with two-way feedback to their care team, all sent by SMS/text message at the participant's preferred time of day. If they indicate that they are in high distress, or they request, their care provider will be notified and asked to reach out to them. They will also receive crisis resources.The intervention will continue until the patient attends the first consultation appointment, or for up to 30 days if the patient does not attend, which reflects the program's practice of closing referrals for non-attending patients.
  Arms: Active SMS Intervention
Behavioral: Sham SMS — Single welcome message letting participant know they will be contacted to book an appointment.
  Arms: Sham SMS

SUMMARY:
Psychosis is a disabling condition that typically has its onset in adolescence and early adulthood. Many young people with psychosis have difficulty navigating services or are reluctant to engage in treatment until their illness becomes an emergency. Consequently, nearly half of all new psychotic disorders are diagnosed in the emergency department (ED). Despite the rationale and evidence for early psychosis intervention (EPI), around half of youth do not access these services. The investigators will use short message service (SMS)/text messaging, a low-cost, low-complexity, youth-friendly approach, to improve transitions in care from the ED and related acute services to EPI services, investigating the intervention's effect on attendance at the first consultation appointment, longer term service engagement, and system-level outcomes. The investigators will also evaluate cost-effectiveness and user perspectives of the intervention.

DETAILED DESCRIPTION:
At the Centre for Addiction and Mental Health (CAMH), the investigators will recruit a consecutive series of 186 participants aged 16 to 29 referred by the CAMH ED and related acute services to CAMH's EPI program for a pragmatic randomized controlled trial of a 2-way SMS intervention involving reminders, psychoeducation, and check-ins. The primary outcome will be rate of attendance at the first consultation appointment assessed through chart reviews. Secondary outcomes will include indicators of long-term service engagement as well as symptoms and functioning 6 months following study enrollment and health service utilization for up to 2 years using administrative data from the Institute for Clinical Evaluative Sciences (ICES). Administrative data will be used for an economic analysis. Participants who receive the active intervention will be asked to complete a web-based survey evaluating their experience and a subgroup will be asked to participate in in-depth in-person qualitative interviews. Patients and family members with lived experience will be engaged in all aspects of the project, including shaping the intervention and study design.

The investigators hypothesize that the intervention will result in increased rate of attendance at the first EPI consultation appointment, as well as improved longer-term engagement in outpatient EPI services compared to the sham comparator. Demonstrating evidence that this low-cost, low-complexity, youth-friendly intervention improves engagement in outpatient EPI services has the potential to improve long-term outcomes for young people with psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Have been referred by the Centre for Addiction and Mental Health (CAMH) emergency department or related acute services to the CAMH early psychosis intervention (EPI) program for suspected psychosis

Exclusion Criteria:

* Inability to communicate in basic written English

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 186 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Attendance at the first early psychosis intervention (EPI) consultation appointment | 30 days
  Attendance at the outpatient EPI consultation appointment will be assessed through chart reviews and categorized as: Yes - attended at original appointment time, Yes - attended at later date within 30 days, No - did not attend appointment within 30 days.

SECONDARY OUTCOMES:
Service engagement - absolute drop-out | 6 months
  Absolute dropouts will be assessed through chart reviews and categorized as: Still in EPI treatment, Not accepted for EPI treatment, Accepted for EPI treatment but transitioned to local services, Accepted for EPI treatment but disengaged, or Other.
Service engagement - Service Engagement Scale (SES) | 6 months
  The Service Engagement Scale is a brief, validated, clinician-rated tool designed to measure engagement with community mental health services. In 14 items, it assesses patients' availability for treatment, collaboration, help seeking behaviors and treatment adherence on a four-point Likert scale with total scores ranging from 0-42, and higher scores indicating difficulties in service engagement. The Service Engagement Scale total score and treatment adherence score will be extracted through chart reviews.
Change in psychotic illness as measured by the Clinical Global Impression (CGI) | 6 months
  The Clinical Global Impression (CGI) is a clinician-rated measure of the patient's symptom severity and treatment response prior to and after initiating an intervention. It includes subscales for Severity and Improvement. The Clinical Global Impression - Severity scale ranges from 1-7 with higher scores indicating higher severity of illness, relative to other patients with the same diagnosis. The Clinical Global Impression - Improvement scale ranges from 1-7 with 4 indicating no change, 1 indicating very much improved, and 7 indicating very much worse relative to the patient's illness at the beginning of the intervention. Scores will be extracted through chart reviews.
System-level outcomes: emergency department visits | 6 months and 2 years
  Number of emergency department visits, extracted from provincial administrative data held at the Institute for Clinical Evaluative Sciences (ICES)
System-level outcomes: mental health hospitalizations | 6 months and 2 years
  Number of mental health hospitalizations, extracted from provincial administrative data held at the Institute for Clinical Evaluative Sciences (ICES)
System-level outcomes: days in mental health hospitalizations | 6 months and 2 years
  Number of days in mental health hospitalizations, extracted from provincial administrative data held at the Institute for Clinical Evaluative Sciences (ICES)
System-level outcomes: outpatient mental health visits with primary care provider | 6 months and 2 years
  Number of outpatient mental health visits with primary care provider, extracted from provincial administrative data held at the Institute for Clinical Evaluative Sciences (ICES)
System-level outcomes: outpatient mental health visits with psychiatrist | 6 months and 2 years
  Number of outpatient mental health visits with psychiatrist, extracted from provincial administrative data held at the Institute for Clinical Evaluative Sciences (ICES)
System-level outcomes: continuous prescriptions | 6 months and 2 years
  For participants with provincial drug coverage, continuous vs. non-continuous prescriptions for antipsychotic or mood stabilizer medications, extracted from provincial administrative data held at the Institute for Clinical Evaluative Sciences (ICES)
System-level outcomes: mortality | 6 months and 2 years
  Mortality, extracted from provincial administrative data held at the Institute for Clinical Evaluative Sciences (ICES)
Health care costs | 6 months and 2 years
  Total direct patient-level health care costs incurred by the public third-party payer based on administrative data held at the Institute for Clinical Evaluative Sciences (ICES) using an established costing algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Kozloff, MD, SM, Principal Investigator — Centre for Addiction and Mental Health; George Foussias, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health; Aristotle N Voineskos, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health; Vicky Stergiopoulos, MD, MHSc, Principal Investigator — Centre for Addiction and Mental Health; Albert HC Wong, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data (IPD) other than system-level data held at ICES will be available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 12 months of posting the study results on this website
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the study's Steering Committee and after Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Polillo A, Foussias G, Wong AHC, Ampofo A, Stergiopoulos V, Anderson KK, Bromley S, D'Arcey J, de Oliveira C, Duda L, Henderson J, Kidd S, Kurdyak P, Wang W, Zaheer J, Voineskos AN, Kozloff N. ED to EPI: protocol for a pragmatic randomised controlled trial of an SMS (text) messaging intervention to improve the transition from the emergency department to early psychosis intervention for young people with psychosis. BMJ Open. 2020 Dec 17;10(12):e042751. doi: 10.1136/bmjopen-2020-042751. PMID 33334839